CLINICAL TRIAL: NCT01103557
Title: The Effectiveness of Prophylactic Selective Lateral Neck Dissection in Papillary Thyroid Carcinoma Patients With Central Neck Metastasis
Brief Title: Prophylactic Selective Lateral Neck Dissection in Patients With Papillary Thyroid Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Yun-Sung Lim, Pusan National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PTC_CND_LND
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-01

CONDITIONS: Thyroid Neoplasm; Lymphatic Metastasis
Keywords: Papillary thyroid carcinoma with neck metastasis; neck dissection
MeSH Terms: conditions — Thyroid Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: prophylactic selective lateral neck dissection — Level II, III, IV lymph node dissection

SUMMARY:
The purpose of this study is to prospectively analyze the incidence of occult lateral neck metastasis (LNM) and to elucidate the factors that predict LNM in papillary thyroid carcinoma (PTC) with central neck metastasis (CNM) by performing prophylactic selective lateral neck dissection (SND).

DETAILED DESCRIPTION:
The lymphatic drainage pattern of the thyroid is uniform and consistent, and therefore, metastatic patterns are relatively predictable. Initial nodal metastasis in PTC usually occurs in the paratracheal and pretracheal nodes in level VI of the central compartment of the ipsilateral neck and spreads to the lateral cervical lymph nodes. Macroscopic skip metastases to the lateral compartment of the neck in the absence of central disease are uncommon.

ELIGIBILITY:
Inclusion Criteria:

* Papillary thyroid carcinoma with central neck metastasis
* No evidence of lateral neck metastasis as determined by high-resolution neck ultrasonography and computed tomography

Exclusion Criteria:

* History of previous thyroid operation
* Isthmic thyroid lesion

Ages: 20 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)